CLINICAL TRIAL: NCT06922955
Title: A Prospective, Open-label, Multi-center, Non-inferiority Study Comparing VivAer® to Alternative Surgical Procedures to Treat Nasal Airway Obstruction in Patients With Nasal Valve Dysfunction (The CompAer Study).
Brief Title: A Prospective Study Comparing VivAer to Alternative Surgical Procedures to Treat Nasal Airway Obstruction in Patients With Nasal Valve Dysfunction.
Acronym: CompAer
Status: Recruiting | Type: Observational
Sponsor: Aerin Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: CTP1563
Record Dates: First submitted 2025-03-26; First posted 2025-04-11 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Nasal Airway Obstruction
Keywords: NAO; Nasal Airway Obstruction; Nasal; Nasal Airway; CompAer; VivAer; nasal valve dysfunction; NOSE
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- VivAer Arm: The VivAer treatment arm will be comprised of patients undergoing the minimally invasive VivAer procedure using the VivAer Stylus and Aerin Console. The VivAer Stylus is a disposable handheld device capable of delivering bipolar radiofrequency (RF) energy to tissue when connected to the Aerin Console radiofrequency generating device. Treatments will be performed using the VivAer Stylus and Aerin Console using non-overlapping and device default settings (temperature 60° C, power 4 watts, treatment time 18 seconds, and cooling time 12 seconds). VivAer treatment areas will include at minimum the lateral nasal wall in the area of the upper lateral cartilage and may also involve treatment of the inferior turbinate and/or septal swell body at the discretion of the investigator according to individual patient needs.
- Surgical Comparator Arm: The two surgical intervention arms will be comprised of patients undergoing surgical intervention for the treatment of NAO as follows:
  * Functional Rhinoplasty Arm: This arm will include patients undergoing primary functional rhinoplasty surgery for NAO addressing the nasal valve and/or lateral nasal wall and may be performed with septoplasty or turbinoplasty performed alone or in combination). This procedure may include minor aspects of cosmesis (e.g., dorsal hump reduction) at the discretion of the investigator.
  * Septoplasty arm: This arm will include patients undergoing a septoplasty with or without turbinate reduction as the only procedures performed for NAO.

SUMMARY:
The purpose of this study is to compare the clinical outcomes of the VivAer procedure to functional rhinoplasty and septoplasty surgery for the treatment of nasal airway obstruction (NAO) to establish non-inferiority.

DETAILED DESCRIPTION:
The purpose of this study is to compare the clinical outcomes of the VivAer procedure to functional rhinoplasty and septoplasty surgery for the treatment of nasal airway obstruction (NAO) to establish non-inferiority by using the NOSE scale to evaluate the significance of a patient's nasal obstruction both before and after the procedure for the primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Age 22 to 85 years old (inclusively).
* Willing and able to provide consent.
* Willing and able to comply with the patient-specific requirements outlined in the study protocol.
* Has access to a mobile device, tablet, or computer with internet access and has access to an email address.
* Seeking treatment for NAO
* Has a NOSE Score of ≥55 indicating severe to extreme NAO.
* Have a positive modified Cottle maneuver.
* Planning either to undergo an intervention for NAO that includes one of the following as the primary approach:

  1. VivAer procedure for repair of nasal valve dysfunction (may include inferior turbinate and septal swell body as additional treated areas)
  2. Functional rhinoplasty surgery addressing the nasal valve and/or lateral nasal wall (may be combined with septoplasty with/without turbinoplasty performed alone or in combination).
  3. Septoplasty surgery with turbinate reduction.

Exclusion Criteria:

* Has had nasal surgery (including sinus surgery) within the last 3 months.
* Has had a previous rhinoplasty (functional or cosmetic), septoplasty, inferior turbinate reduction, or VivAer procedure.
* Has extreme nasal pathology, a history of extreme nasal injuries, or an abnormal nasal condition (e.g. septal perforation or empty nose syndrome) that may be exacerbated by surgery.
* Has a medical condition(s) that may impair normal healing processes or be exacerbated by the stress of surgery.
* Has chronic rhinitis that is refractory to medications or rhinitis medicamentosa.
* Has poorly controlled chronic rhinosinusitis disease.
* Rhinoplasty is being performed primarily for cosmesis.
* Is receiving, planning to receive, or has received a Latera absorbable nasal implant at any time.
* Planning to have sinus or cosmetic surgery (e.g., functional endoscopic sinus surgery, cosmetic rhinoplasty) or a surgery involving the airway (e.g., hypoglossal nerve stimulation surgery, uvuloplasty, tonsillectomy, tongue base or soft palate interventions) within 6 months following enrollment.
* Is having an adjunctive surgical procedure performed with the primary NAO procedure (e.g. functional rhinoplasty with concha bullosa reduction, septoplasty with turbinate reduction performed with functional endoscopic sinus surgery)

Ages: 22 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 22-85 seeking treatments for nasal airway obstruction.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Nasal Obstruction Symptom Evaluation (NOSE) Scale | 3 months, 6 months, 12 months and 24 months post-procedure.
  To evaluate the significance of a patient's nasal obstruction both before and after the procedure for the primary endpoint, this study will use the well-known subjective patient-reported outcome measure, the NOSE Scale. The NOSE Scale is a validated disease-specific health status instrument used by clinicians to measure outcomes of participants treated for nasal obstruction. The NOSE Scale consists of 5 items, each scored using a 5-point Likert scale with a total score range of 0 through 100, where higher scores indicate worse obstruction. Severity of symptoms can be classified as mild (range, 5-25), moderate (range, 30-50), severe (range, 55-75), or extreme (range, 80-100) nasal obstruction, based on responses to the NOSE survey.
  Individual participant success (treatment responder) is based on NOSE Scale improvement defined as a ≥ 24 point improvement (decrease) in NOSE Scale score from baseline to the 3-month evaluation.

SECONDARY OUTCOMES:
Epworth Sleepiness Scale (ESS) | 3 months, 6 months, 12 months and 24 months post-procedure.
  The ESS evaluates the self-reported likelihood of dozing or falling asleep in 8 daytime situations with likelihood rated as No Chance (0), Slight (1), Moderate (2), or High Chance (3).
12-item Short Form (SF-12) Survey | 3 months, 6 months, 12 months and 24 months post-procedure.
  The SF-12 is one of the most widely used instruments for assessing self-reported health-related quality of life, and has been validated in numerous studies.40 The SF-12 is a general health questionnaire that consists of 12 questions which investigates the patient's perception about their state of health via 8 different dimensions: General health perception - 1 question, Physical health - 2 questions, Limited physical role function - 2 questions, Physical pain - 1 question, Vitality - 1 question, Mental health - 2 questions, Limited emotional role function - 2 questions, and Social functioning - 1 question. Two summary scores are reported from the SF-12 - a mental component score (MCS-12) and a physical component score (PCS-12). Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning. A score above 50 indicates better than average health-related quality of life and scores less than 50 suggest below-average health.41
Visual Analogy Scale (VAS) Score | 1 week post procedure
  The Visual Analogue Scale (VAS) is a unidimensional measure of pain intensity that will be used to measure nasal pain associated with the procedure.39 A VAS is usually a 100-mm long horizontal line with verbal descriptors (word anchors) at each end to express the extremes of the feeling. Scores are obtained by measuring the distance in millimeters from the left origin of the line (0) to the point indicated with a slash placed by the patient to indicate their current level of pain in and around the nose. Results are then assigned a score between 0 and 100.
Return to Work | 3 months post procedure.
  Assessment of the number of workdays missed within the first month due to the receiving the procedure will be collected.
Patient Satisfaction with Procedure | 3 months, 6 months, 12 months and 24 months post-procedure.
  Satisfaction with the procedure is measured with a five-question, self-reported survey using a 5-point scale to assess tolerability of the procedure, ease of recovery, change in NAO symptoms, overall satisfaction with the procedure, and recommendation to others.
Adverse Events | Through study completion, minimum 2 years
  Physician and patient reported adverse events will be collected.

CONTACTS AND LOCATIONS:
Locations (35):
- United States (35):
  - Southern Head and Neck Surgery, Alexander City, Alabama
  - ExcelENT, Birmingham, Alabama
  - North Alabama ENT, Huntsville, Alabama
  - East Alabama ENT, Opelika, Alabama
  - Arizona Desert ENT Specialists, Goodyear, Arizona
  - Honor Health ENT, Scottsdale, Arizona
  - Tucson ENT, Tucson, Arizona
  - Cedars Sinai Medical Center, Los Angeles, California
  - Alexis Furze, MD Inc, Newport Beach, California
  - Sacramento ENT (DaVinci Research), Roseville, California
  - Mercy Medical Group, Sacramento, California
  - Breathe Clear Institute, Torrance, California
  - IMMUNOe Research Center, Denver, Colorado
  - ENT & Allergy Associates of Florida (Boynton Beach), Boynton Beach, Florida
  - Advanced ENT and Allergy, Fernandina Beach, Florida
  - ENT and Allergy Associates of Florida, Plantation, Florida
  - ENT and Allergy Associates Of Florida, Port Saint Lucie, Florida
  - ENT and Allergy Associates of Florida (West Palm Beach), West Palm Beach, Florida
  - Chicago Nasal and Sinus Center, Chicago, Illinois
  - Chicago ENT, Chicago, Illinois
  - Kentuckia Ear Nose & Throat, Louisville, Kentucky
  - Dearborn ENT, Dearborn, Michigan
  - Dearborn ENT Livonia, Livonia, Michigan
  - Maddison ENT, New York, New York
  - Madison ENT, New York, New York
  - Open Sinus, New York, New York
  - University of Rochester, Rochester, New York
  - Bethlehem ENT /Specialty Physician Associates, Bethlehem, Pennsylvania
  - ENT Associates of Texas, McKinney, Texas
  - Hill Country ENT, New Braunfels, Texas
  - Endormir Sleep Solution LLC, San Antonio, Texas
  - Texas Facial Plastic Surgery & ENT, San Antonio, Texas
  - Alamo ENT Associates, San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia
  - ENT & Allergy Associates, Puyallup, Washington

IPD SHARING:
Plan to Share IPD: No